CLINICAL TRIAL: NCT02838797
Title: RQ-00000010 for Gastroparesis and Constipation in Parkinson's Disease
Acronym: RQ-10
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); RaQualia Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20001657
Record Dates: First submitted 2016-06-16; First posted 2016-07-20 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Parkinson's Disease; Gastroparesis; Constipation
Keywords: Parkinson's disease; Gastroparesis; Constipation; Prokinetic; 5-HT4-receptor partial agonist
MeSH Terms: conditions — Parkinson Disease; Gastroparesis; Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): For the single ascending dose study, subjects will receive a single dose of oral acetate buffer on a single day.
  For the multiple ascending dose study, subjects will receive a single daily dose of oral acetate buffer each day for 14 days.
  Interventions: Drug: Placebo
- RQ-00000010 (Experimental): For the single ascending dose study, subjects will receive a single dose of either:
  2 micrograms, 50 micrograms or 200 micrograms of RQ-00000010 on a single day.
  For the multiple ascending dose study, subjects will receive single daily doses of either 10 micrograms, 50 micrograms or 100 vs. 200 micrograms of RQ-00000010 each day for 14 days.
  Interventions: Drug: RQ-00000010

INTERVENTIONS:
Drug: RQ-00000010 — orally administered serotonin 4 receptor partial agonist
  Arms: RQ-00000010
Drug: Placebo — oral acetate buffer
  Arms: Placebo

SUMMARY:
This is a study to determine the safety and tolerability of a new medicine (RQ10) for gastrointestinal symptoms in Parkinson's disease. The investigators will also begin to look at the effect of this medicine on gastrointestinal problems. The results will determine if future studies are appropriate. In this study, RQ10 will be compared to a placebo (a look-alike inactive substance). Participation will include multiple office visits. Approximately 48 people will participate.

DETAILED DESCRIPTION:
This is a phase Ib study with the primary objectives of determining the safety and tolerability as well as pharmacokinetics after single ascending doses (SAD) and multiple ascending doses (MAD) of RQ10 in Parkinson's disease patients. A secondary objective will be to assess the impact of single doses of RQ10 on gastric emptying in Parkinson's Disease patients as well as the effects of RQ10 on gastroparesis symptoms. The expected results of this exploratory phase Ib study will allow deciding about whether to proceed with further development of RQ10 in Parkinson's Disease patients ("go-no go") and help design a formal phase IIa "proof of concept" study by informing repeat-dose selection and possible effect sizes in Parkinson's Disease patients.

ELIGIBILITY:
Inclusion Criteria: For both the Single Ascending Dose and Multiple Ascending Dose studies: Idiopathic Parkinson's Disease (UK Brain Bank Criteria), Hoehn & Yahr stages 1-3, participants may be on oral levodopa, dopamine agonists, monoamine oxidase-B inhibitors, catechol-O-methyltransferase inhibitors, and amantadine, but doses must have remained stable for 28 days prior to enrollment and should be anticipated to remain stable throughout the study, participants may have deep brain stimulation (though stimulator settings must be expected to remain constant throughout the study) or ablative surgery for Parkinson's Disease.

Additional Inclusion criteria for the Multiple Ascending Dose study only: Must have symptoms suggestive of current gastroparesis or constipation as shown by any one or more of the following: 1. Need for regular use of prokinetics, laxatives, or stool softeners of any kind, 2. A total score of 2 or higher on the Gastroparesis Cardinal Symptoms Index (total score equals average of scores on the 3 subscales), 3. A score of 5 or higher on the gastroparesis subscale or 5 or higher on the constipation subscale of the Gastrointestinal Symptoms in Neurodegenerative Disease Scale.

-

Exclusion Criteria: Dementia (Mini Mental Status Exam < 25), active psychosis, severe depression (score of 4 on question 1.3 of the Movement Disorder Society-United Parkinson Disease Rating Scale), active suicidality as measured by a most severe suicide ideation score of 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS), or patients who answer "Yes" on any of the 5 C-SSRS Suicidal Behavior Items if the attempt or acts were performed within 1 year of screening, or patients who, in the opinion of the investigator, present a risk of suicide, any chronic gastrointestinal diseases except gastroesophageal reflux disease, history of any gastrointestinal surgery that might impact drug absorption (e.g. gastrectomy), use of apomorphine, anticholinergics, or carbidopa/levodopa intestinal gel for Parkinson's Disease, female participants who are pregnant or lactating, male or female participants of childbearing age who are not willing, or whose partners are not willing, to use contraception during the study, diabetes, symptomatic anemia, abnormal liver or kidney function, cardiac arrhythmia (past or present) or abnormal QT interval on entrance electrocardiogram, positive drug screen at screening visit, allergy to spirulina, egg, milk, or wheat, pulmonary dysfunction (e.g. Chronic Obstructive Pulmonary Disease), small bowel malabsorption, use of any medications affecting gastric emptying (macrolides, metoclopramide, domperidone, opiates, anticholinergics) within 3 days of visits 2 and 3, prisoners, and individuals with limited English proficiency.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 18 months
  adverse events, serious adverse events, electrocardiograms, physical exams, vital signs and safety labs

SECONDARY OUTCOMES:
Gastric emptying | 1 hour after RQ10 dosing
  Carbon 13 Breath Test kit by Cairn Diagnostics
Area Under the Curve [AUC] for RQ-00000010 after single and multiple doses | 18 months
Peak Plasma Concentration (Cmax) for RQ-00000010 after single and multiple doses | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Cloud, MD, MSc, Principal Investigator — Virginia Commonwealth University
Locations (1):
- VCU NOW Center, Henrico, Virginia, United States